CLINICAL TRIAL: NCT03648424
Title: Prediction of Findings From the Ongoing CAROLINA Trial Using Healthcare Database Analyses
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elisabetta Patorno, Assistant Professor of Medicine at Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: 2013P002157
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Linagliptin; Cardiovascular Death; Stroke; Myocardial Infarction; Hospitalization for Unstable Angina; Type 2 diabetes mellitus; Glimepiride
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Stroke; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Linagliptin: Patients who initiate Linagliptin with no use in the prior 180 days
- Glimepiride: Patients who initiate Glimepiride with no use in the prior 180 days

SUMMARY:
This cohort study was initiated to predict the findings of CAROLINA trial in a real world setting using electronic claims data from insurance databases with results anticipated prior to the completion of CAROLINA.

DETAILED DESCRIPTION:
The CARdiovascular Outcome Trial of LINAgliptin Versus Glimepiride in Type 2 Diabetes (CAROLINA) is an ongoing randomized controlled trial (RCT) designed to assess whether linagliptin is non-inferior, and if so, superior compared with glimepiride 1-4 mg once daily with respect to cardiovascular (CV) events in adults with relatively early Type 2 Diabetes at increased risk of CV events and with less than optimized glycaemic control. Given that medications of both classes are currently advocated as second-line therapy after metformin, and since sulfonylureas have been associated with concerns regarding their CV safety, while dipeptidyl peptidase-4 inhibitors have been suggested to exhibit CV benefits in preclinical and mechanistic trials, the results of this trial will provide answers to several clinically relevant questions and have a significant impact on clinical practice.

This cohort study was initiated to predict the findings of CAROLINA trial in a real world setting using electronic claims data from insurance databases with results anticipated prior to the completion of CAROLINA. Trial eligibility criteria were adapted in claims data to generate a comparable study cohort (of linagliptin and glimepiride initiators) to that of the trial population. Using 1:1 propensity score-matching was used to control for >120 baseline characteristics. Patients were followed up for a composite cardiovascular outcome adapted from the primary end-point of the CAROLINA trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes who were new users of Linagliptin or new users of Glimepiride and:

  - Had no more than 3 anti-diabetic drugs including index drug
* AND at elevated risk of cardiovascular (CV) events according to specific criteria:

  * Previous vascular disease
  * Evidence of vascular-related end-organ damage
  * Age ⩾ 70 years
  * ⩾ 2 CV risk factors:

    * Treated hypertension
    * Smoking
    * Using any lipid lowering treatment
* Age ≥ 40 and ≤ 85 years at treatment initiation

Exclusion Criteria:

* Patients with Type 1 Diabetes Mellitus
* Previous exposure to dipeptidyl peptidase-4 (DPP-4) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists, thiazolidinediones (TZDs), insulin or sodium glucose co-transporter-2 (SGLT-2s).
* Exclude anti-diabetic background therapy if initiated in 2 months prior
* Morbid obesity or treatment with anti-obesity drugs 3 months prior to treatment initiation
* Severe hyperglycemia
* Active liver disease or impaired hepatic function
* Any previous bariatric surgery
* Coronary artery re-vascularisation ≤ 6 weeks prior to treatment initiation
* Prior hospitalization for congestive heart failure
* Acute or chronic metabolic acidosis
* Hereditary galactose intolerance
* Alcohol or drug abuse within the 3 months prior to treatment initiation
* Use of oral corticosteroids
* Pregnant women
* Patients with cancer
* Acute coronary syndrome ≤ 6 weeks prior to treatment initiation
* Stroke or Transient ischemic attack ≤ 3 months prior to treatment initiation

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 40 - 85 years of age with early Type 2 Diabetes mellitus, increased cardiovascular risk or established complications
Sampling Method: Non-Probability Sample
Enrollment: 48262 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Composite Cardiovascular (CV) Outcome | From treatment initiation to end of follow-up, up to 53 months
  Composite CV Outcome includes Myocardial infarction, Stroke, hospitalization for unstable angina and Death

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Patorno, MD DrPH, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Patorno E, Schneeweiss S, Gopalakrishnan C, Martin D, Franklin JM. Using Real-World Data to Predict Findings of an Ongoing Phase IV Cardiovascular Outcome Trial: Cardiovascular Safety of Linagliptin Versus Glimepiride. Diabetes Care. 2019 Dec;42(12):2204-2210. doi: 10.2337/dc19-0069. Epub 2019 Jun 25. PMID 31239281
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727